CLINICAL TRIAL: NCT03378765
Title: Gut Microbiota, Short Chain Fatty Acids, and Adiposity Across The Epidemiological Transition
Status: Active, not recruiting | Type: Observational
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Lara Dugas, Assistant Professor, Loyola University
Other Study IDs: 209537
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- African origin adults: African origin adults from Ghana, Jamaica, Seychelles, South Africa and USA between the ages of 30- 50.
  Interventions: Behavioral: Diet and physical activity monitoring

INTERVENTIONS:
Behavioral: Diet and physical activity monitoring — Lifestyle monitoring

SUMMARY:
The objective of this study is to define associations between gut microbiota, SCFAs and obesity in populations spanning the epidemiologic transition, and explore mechanisms by which these factors may independently and collectively influence the development of obesity. The central hypothesis of this study is that the composition of gut microbiota drives SCFA production which in turn influences obesity risk at the population-level.

DETAILED DESCRIPTION:
The objective of this study is to define associations between gut microbiota, short chain fatty acids (SCFAs) and obesity in populations spanning the epidemiologic transition, and explore mechanisms by which these factors may independently and collectively influence the development of obesity. The gut microbiota and SCFAs have been associated with obesity, yet the causal mechanisms are unknown, as are the individual obesogenic effects of the individual SCFAs (butyrate, acetate and propionate). Existing studies are, limited by contradictory findings, small sample sizes, limited and imprecise measurements of obesity, and lack of detailed dietary and other environmental exposures/mediators. The investigators propose to overcome these challenges by leveraging an existing cohort of five diverse, well-defined populations from the Modeling the Epidemiologic Transition Study (METS, R01-DK080763). METS is comprised of a cohort of 2,500 African-origin adults, living in 5 distinctly different environments; Ghana, South Africa, Jamaica, the Seychelles and the US, and who have been prospectively followed since 2010. Our preliminary data suggest that while gut microbiota and SCFAs differences exist across sites, similar relationships exist across the sites for gut microbiota/SCFAs adiposity effects. In addition to yearly health measurements; the investigators propose to measure gut microbiota and stool SCFAs in all participants (2500) during the first year of the current study, thus providing one of the largest gut microbiota population-based studies to date. We will divide our cohort of 2500 individuals into 2 sets: (1) a test set of 1000 participants to explore which gut microorganisms and stool SCFAs are associated with adiposity; (2) a validation set of 1500 participants to independently verify the biomarkers identified in the test set, thus minimizing spurious correlations due to large number of features (e.g., bacterial taxa). The investigators will follow all 2500 participants for 3 years to assess weight and adiposity changes, using Bayesian Kernel Machine Regression modeling to explore whether changes can be predicted by gut microbiota and SCFAs factors. Finally, using a causal mediation analysis, the investigators will identify the direct and indirect effect of single and/or cumulative gut microbiota on adiposity as mediated by SCFA. The investigators will thus capitalize upon an existing, extensively well described cohort of adults of African-origin, with significant variability as a result of the widespread geographic distributions, and therefore variation in the environmental covariate exposures. The proposed study will substantially advance the understanding of the role gut microbiota and SCFAs play in the development of obesity and provide novel obesity therapeutic targets targeting SCFAs producing features of the gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Identify as African American or Black
* Age 18-50

Exclusion Criteria:

* Pregnancy, nursing, or planning to become pregnant
* Movement disorders or other disability that limits mobility

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study is comprises a complex samples population based approach drawn from communities in 5 countries: Ghana, Seychelles, South Africa, Jamaica and the US. Approximately 500 participants are enrolled per site for an unweighted total of 2500 participants.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
BMI | 24 months
  Difference in body weight index (BMI) between high and low activity energy expenditure (AEE) groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Chicago, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luke A, Bovet P, Forrester TE, Lambert EV, Plange-Rhule J, Schoeller DA, Dugas LR, Durazo-Arvizu RA, Shoham D, Cooper RS, Brage S, Ekelund U, Steyn NP. Protocol for the modeling the epidemiologic transition study: a longitudinal observational study of energy balance and change in body weight, diabetes and cardiovascular disease risk. BMC Public Health. 2011 Dec 14;11:927. doi: 10.1186/1471-2458-11-927. PMID 22168992
- [Derived] Dugas LR, Lie L, Plange-Rhule J, Bedu-Addo K, Bovet P, Lambert EV, Forrester TE, Luke A, Gilbert JA, Layden BT. Gut microbiota, short chain fatty acids, and obesity across the epidemiologic transition: the METS-Microbiome study protocol. BMC Public Health. 2018 Aug 6;18(1):978. doi: 10.1186/s12889-018-5879-6. PMID 30081857
- See also: METS microbiome project website — https://ssom.luc.edu/public_health_sciences/researchprograms/currentresearchprograms/gutmicrobiotashortchainfattyacidsadiposity/